CLINICAL TRIAL: NCT04128592
Title: Non-invasive Differential Diagnosis of Noisy Breathing Infants and Toddlers Based on Biomarker Profiles in Exhaled Breath and Nasal Mucus and Based on Breath Sound Analysis
Brief Title: Non-invasive Differential Diagnosis of Noisy Breathing Infants and Toddlers
Acronym: NiNbI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); VITO (Unknown)
Responsible Party: Principal Investigator, Marc Raes, prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NiNbI-001
Record Dates: First submitted 2019-08-27; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Noisy Breathing Infants; Noist Breathing Toddlers; Wheezing; Rattling
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheezing (Other)
  Interventions: Device: diagnosing noisy breathing in infants and toddlers
- Rattling (Other)
  Interventions: Device: diagnosing noisy breathing in infants and toddlers

INTERVENTIONS:
Device: diagnosing noisy breathing in infants and toddlers — breath sampling and nasal mucus sampling to analyze biomarkers and breath sound analysis to diagnose noisy breathing.

SUMMARY:
Almost 50% of all children have at least 1 episode of noisy breathing before the age of 2 years and almost 25% of these children have more episodes of noisy breathing. The lack of an objective technique for diagnosing noisy breathing children often leads to overrated diagnosis of "wheezing", whereas there may be other noisy breathing phenotypes, like "rattling", that don't favor from the same therapeutic treatment. Presumably, different underlying pathophysiological mechanisms are involved with different biomarker profiles characteristic for different phenotypes. The goal of this study is to optimize the diagnosis of noisy breathing infants and toddlers. Children will be followed for a treatment period of 6 weeks and will visit the paediatrician 3 times (week 0, 3 and 6). During the consultations breath sound analysis will be performed and a breath sample and a nasal mucus will be collected to analyse biomarker profiles. Both methods for diagnosing noisy breathing infants are non-invasive and will be compared to the standard procedure of the paediatrician which consists of auscultation and palpation of the chest. An objective and non-invasive method for diagnosing noisy breathing infants and toddler will pave the way for more cost-effective and personalized prescription of therapies which will increase the quality of life of children with noisy breathing.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of noisy breathing ("wheezing" or "rattling")

Exclusion Criteria:

* born before pregnancy week 37
* congenital or genetic conditions (Down syndrome, Klinefelter's syndrome, …)
* acquired chronic respiratory diseases (bronchopulmonary dysplasy, lung fibrosis, …)

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Noisy breathing diagnosis made by pediatrician based on anamnesis and auscultation | week 0
  Noisy breathing diagnosis is made by the same pediatrician and is based on intensity and duration of both wheeze and rattle are scored on a scale of 0 to 10, whit 0 indicating not present and 10 indicating very high intensity or of continuous duration.
Noisy breathing diagnosis made by pediatrician based on anamnesis and auscultation | week 3
  Noisy breathing diagnosis is made by the same pediatrician and is based on intensity and duration of both wheeze and rattle are scored on a scale of 0 to 10, whit 0 indicating not present and 10 indicating very high intensity or of continuous duration.which differentiate "wheezing" and "rattling" infants and toddlers. Comparing diagnosis based on these biomarker profiles to the diagnosis made by the pediatrician based on auscultation and palpation.
Noisy breathing diagnosis made by pediatrician based on anamnesis and auscultation | Week 6
  Noisy breathing diagnosis is made by the same pediatrician and is based on intensity and duration of both wheeze and rattle are scored on a scale of 0 to 10, whit 0 indicating not present and 10 indicating very high intensity or of continuous duration.which differentiate "wheezing" and "rattling" infants and toddlers. Comparing diagnosis based on these biomarker profiles to the diagnosis made by the pediatrician based on auscultation and palpation.
exhaled breath volatiles | week 0
  exhaled breath volatiles analyzed with Selected Ion Flow Tube Mass Spectrometry (SIFT-MS) and Gas Chromatography Mass Spectrometry (GC-MS)
exhaled breath volatiles | week 3
  exhaled breath volatiles analyzed with Selected Ion Flow Tube Mass Spectrometry (SIFT-MS) and Gas Chromatography Mass Spectrometry (GC-MS)
exhaled breath volatiles | week 6
  exhaled breath volatiles analyzed with Selected Ion Flow Tube Mass Spectrometry (SIFT-MS) and Gas Chromatography Mass Spectrometry (GC-MS)
respiratory pathogens | week 0
  respiratory pathogens present in a nasopharyngeal swab detected using PCR
respiratory pathogens | week 3
  respiratory pathogens present in a nasopharyngeal swab detected using PCR
respiratory pathogens | week 6
  respiratory pathogens present in a nasopharyngeal swab detected using PCR
level of inflammation markers | week 0
  level of inflammation markers in the nasopharyngeal swab using multiplex immune-assay
level of inflammation markers | week 3
  level of inflammation markers in the nasopharyngeal swab using multiplex immune-assay
level of inflammation markers | week 6
  level of inflammation markers in the nasopharyngeal swab using multiplex immune-assay

SECONDARY OUTCOMES:
Breath sound recordings evaluated by expert panel of pediatricians | week 0
  Intensity and duration of both wheeze and rattle are scored on a scale of 0 to 10, whit 0 indicating not present and 10 indicating very high intensity or continuous over the recording.
Breath sound recordings evaluated by expert panel of pediatricians | week 3
  Intensity and duration of both wheeze and rattle are scored on a scale of 0 to 10, whit 0 indicating not present and 10 indicating very high intensity or continuous over the recording.
Breath sound recordings evaluated by expert panel of pediatricians | week 6
  Intensity and duration of both wheeze and rattle are scored on a scale of 0 to 10, whit 0 indicating not present and 10 indicating very high intensity or continuous over the recording.
Treatment response assessed by online journal for parents | week 6
  Parents are asked what type of noisy breathing symptoms their child had during the day. Options are: (1) Wheezing; (2) Rattling; (3) Both, but mostly wheezing; (4) Both, but mostly rattling; (5) Both in equal amounts, (6) No noisy breathing today. In the online questionnaire sound fragments of wheezing and rattling are available incase parents are in doubt.
Recurrence of symptoms assessed by follow up questionnaire | 3 months after week 6
  Online questionnaire asks about noisy breathing symptoms in the past 3 months, their frequency and seriousness. In the online
Recurrence of symptoms assessed by follow up questionnaire | 6 months after week 6
  Online questionnaire asks about noisy breathing symptoms in the past 3 months, their frequency and seriousness. In the online
Recurrence of symptoms assessed by follow up questionnaire | 9 months after week 6
  Online questionnaire asks about noisy breathing symptoms in the past 3 months, their frequency and seriousness. In the online
Recurrence of symptoms assessed by follow up questionnaire | 12 months after week 6
  Online questionnaire asks about noisy breathing symptoms in the past 3 months, their frequency and seriousness. In the online

CONTACTS AND LOCATIONS:
Overall Officials: Marc Raes, prof. dr., Principal Investigator — Jessa Hospital; Gitte Slingers, drs., Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided